CLINICAL TRIAL: NCT02162082
Title: Coronary and Structural Interventions Ulm - Coronary Chronic Total Occlusions
Acronym: CSI-Ulm-CTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Jochen Wohrle, Prof. Dr. Jochen Wöhrle, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI Ulm - CTO 1.0
Record Dates: First submitted 2014-06-07; First posted 2014-06-12 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Stable Angina
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Angina, Stable | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stent or scaffold (Experimental): implantation of stents or scaffolds after recanalization of coronary chronic total occlusions
  Interventions: Device: stent or scaffold

INTERVENTIONS:
Device: stent or scaffold — implantation of a CE certified drug-eluting stent, bare-metal stent or scaffold

SUMMARY:
To evaluate the long-term results after recanalization of coronary chronic total occlusions.

DETAILED DESCRIPTION:
Patients with successful recanalization of coronary chronic total occlusions are followed during a period of 5 years to demonstrate safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease
* chronic total occlusion

Exclusion Criteria:

* no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2014-06; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 1-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wöhrle, MD, Principal Investigator — University of Ulm, Ulm, Germany
Locations (1):
- University of Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kugler C, Markovic S, Rottbauer W, Wohrle J. Bioresorbable scaffolds compared with everolimus-eluting stents for the treatment of chronic coronary total occlusion: clinical and angiographic results of a matched paired comparison. Coron Artery Dis. 2017 Mar;28(2):120-125. doi: 10.1097/MCA.0000000000000449. PMID 27845998